CLINICAL TRIAL: NCT06722560
Title: SHORT-term Effects of GLucagon-like Peptide One on BonE
Acronym: SHORT-GLOBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: S--20240027
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-01

CONDITIONS: To Investigate the Physiological Effect of GLP-1 on the Skeleton; Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLP-1 hormone (Active Comparator)
  Interventions: Other: GLP-1 hormone
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: GLP-1 hormone — s.c. continuous infusion for 72 hours using an insulin pump
  Arms: GLP-1 hormone
Other: Placebo — s.c. continuous infusion for 72 hours using an insulin pump
  Arms: Placebo

SUMMARY:
Bone is a dynamic organ that is remodelled throughout life by a coupled process of resorption and formation of bone tissue, which are highly energy-demanding processes. Bone remodelling is tightly regulated by several endocrine factors such as parathyroid hormone, sex steroids including testosteron and oestrogen, and growth hormone. More recently, gut secreted hormones have emerged as regulators of bone resorption and formation. Glucagon-like peptide 1 (GLP-1) is secreted from the gut following food intake and increases insulin secretion and satiety. Physiological infusion studies using native GLP-1 as subcutaneous or intravenous infusions demonstrate that native GLP-1 maintains bone formation in humans but decreases bone resorption (assessed using the C-terminal telopeptide of type-I collagen (CTX) biomarker) in some but not all studies. The investigators speculate that native GLP-1 signals the presence of nutrients needed for bone expansion of bone mass. The investigators recently extended current knowledge on GLP-1 biology by showing that short-term (2 hours) in-travenous exposure to native GLP-1 (7-36)), the active form of GLP-1, leads to an 80 % reduction in bone resorption based on measures of CTX in the bone marrow in healthy study participants. Our three-day in-vitro experiment based on human bone cells demonstrated that native GLP-1 (7-36) enhances the activity of bone resorbing cells (osteoclasts) and bone forming cells (osteoblasts) when they are cultured together. Jointly, these findings indicate that GLP-1 (7-36) regulates bone cell activi-ty in a time-dependent manner: Within 2 hours, native GLP-1 (7-36) decreases bone resorption but maintains bone formation. By contrast, extended exposure to native GLP-1 (7-36) appears to activate both bone resorbing and forming cells. Importantly, these latter in vitro-based findings have not been corroborated by physiological studies. However, such a time dependent skeletal impact of GLP-1 would be in keeping with the biology of several hormones.

The aim of this study is to investigate the physiological effect of GLP-1 on the skeleton. While there is evidence supporting that GLP-1 regulates bone turnover, the differential effects of acute and extended (sub-acute) exposure to GLP-1 on bone turnover remain to be explored. Therefore, this study aims to elucidate how native GLP-1(7-36) regulates bone formation and resorption in healthy men and women, thus providing further insights into the effects of native GLP-1 (7-36) on human bone metabolism.

This is a randomized crossover study that compares the biological effects of native GLP-1 (7-36) or saline on bone formation in 12 healthy individuals. The study consists of an information visit, a screening visit with a general health assessment and four experimental days. Native GLP-1 (7-36) (1 pmol/kg/min) or saline will be administered subcutaneous using a commercially available insulin pump for 72 hours with a wash-out period of 14-28 days between exposures. The sequence of exposure is randomized, and the participants are blinded.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Diabetes mellitus including prediabetes (Hb1Ac >42 mmol/mol at baseline)
* BMI > 28 kg/m2
* Conditions and pharmaceutical treatments that influence bone metabolism (e.g., bone fractures < 6 months, uncontrolled thyrotoxicosis, and severe renal impairment).
* Pregnancy
* Inability to complete all investigations or to provide informed consent

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Change in serum bone formation marker P1NP | Between baseline and day 4

SECONDARY OUTCOMES:
Change in serum bone resorption marker CTX | Between baseline and day 4, compared with baseline results.
Serum levels of GLP-1 | Between baseline and day 4

OTHER OUTCOMES:
Bone turnover markers P1NP and CTX in bone marrow serum | Between baseline and day 4

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology, University Hospital of Odense, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No